CLINICAL TRIAL: NCT02904083
Title: Study of the Effectiveness of Specific Training of Health Professionals on Adherence in Bipolar Disorder
Acronym: CONCORDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2015-07
Record Dates: First submitted 2016-09-08; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Bipolar Disorders
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- specific training of professionals (Experimental): patients from centers where professionals have received specific training
  Interventions: Behavioral: self assessment of adherence
- control training of professionals (Active Comparator): patients from centers where professionals have received control training
  Interventions: Behavioral: self assessment of adherence

INTERVENTIONS:
Behavioral: self assessment of adherence

SUMMARY:
Bipolar disorders are common psychiatric disorders characterized by severe and recurrent symptomatic periods (Major Depressive Episode, mania, hypomania) and interictal periods characterized by persistent residual symptoms, impaired functioning and quality of life. In addition, the prognosis of bipolar disorder is aggravated by an increased risk of suicide and a high frequency of somatic comorbidities. Poor adherence is one of the major factors influencing the course of the disorder and one of the causes of ineffective treatments. Considering that between 20 and 60% of patients with bipolar disorder have problems with adherence. Adherence is modulated by a number of socio-demographic, clinical and neuropsychological factors. It is also modulated by the knowledge, beliefs and In addition, studies have shown that the reasons attributed to poor adherence are different depending on whether questioning patients or healthcare professionals. This fault diagnosis, assessment of the causes and "fit" into the reasons associated with poor adherence is an aggravating factor of the problem. However, this factor seems modifiable by better training of professionals. A team from Newcastle University in England has developed a training program for all health professionals to improve the diagnosis and understanding of compliance issues in bipolar patients and provide simple tools to fight against patients with this problem. The investigators assume that this training will improve medication adherence among outpatients by trained professionals.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from bipolar disorder type 1, type 2 or unspecified according to the DSM IV
* Do not presenting mood episode as defined in DSM IV
* With at least one medication prescribed mood stabilizer goal, whatever its observance

Exclusion Criteria:

* Patients full-time hospitalized at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-06; Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Difference of score of Medication Adherence Rating Scale (MARS) before and after the training of the professionals | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No